CLINICAL TRIAL: NCT01176617
Title: Assessment of Arrhythmia Burden in Patients Undergoing Atrial Fibrillation Using an Implantable Loop Recorder (ILR) Versus Conventional Monitoring Strategy
Brief Title: Assessing Arrhythmias After Ablation Using Implantable Recorders
Acronym: ABACUS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UPenn811675
Record Dates: First submitted 2010-08-04; First posted 2010-08-06 (Estimated); Results first posted 2018-04-05 (Actual); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation; A-Fib; AF; Persistent; Permanent; Pulmonary Vein isolation; Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional Monitoring Strategy (No Intervention): Subjects will be monitored for 12 months using the conventional strategy which includes wearing a monitor over 3 separate 30-day periods over the first year post-ablation and daily pulse checks.
- Reveal XT (Other): Subjects will be monitored using the conventional monitoring strategy for the first 6 months post-ablation. During the next 6 months, subjects will be monitored using the data from the Reveal device, transmitted from home every 30 days.
  Interventions: Device: Reveal XT implantable loop recorder

INTERVENTIONS:
Device: Reveal XT implantable loop recorder — All study participants will receive the Reveal XT implantable loop recorder immediately after completion of the ablation procedure.
  Arms: Reveal XT

SUMMARY:
The purpose of this study is to determine if continuous monitoring using an implantable loop recorder (ie. a device that is placed just underneath the skin of the chest and monitors the heart rate and rhythm) for a year long period after atrial fibrillation ablation may be superior to the current conventional monitoring strategy used by us for determination of atrial fibrillation recurrence (ie. return of the abnormal heart rhythm) and/or arrythmia burden (ie. how long the abnormal rhythm continues or how often the rhythm occurs). Some data suggests that continuous monitoring over longer periods may be better in identifying recurrence of atrial fibrillation after ablation and thus assist in its overall management. The device being used for this study is the Reveal XT, which, is currently FDA approved for monitoring all varieties of cardiac rhythm disorders including atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years
* Undergoing ablation for atrial fibrillation at the University of Pennsylvania

Exclusion Criteria:

* Patients with already implanted devices, including pacemakers, implantable cardiac defibrillators and cardiac resynchronization devices

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2012-06; Primary Completion 2012-08 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjay Dixit, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Kapa S, Epstein AE, Callans DJ, Garcia FC, Lin D, Bala R, Riley MP, Hutchinson MD, Gerstenfeld EP, Tzou W, Marchlinski FE, Frankel DS, Cooper JM, Supple G, Deo R, Verdino RJ, Patel VV, Dixit S. Assessing arrhythmia burden after catheter ablation of atrial fibrillation using an implantable loop recorder: the ABACUS study. J Cardiovasc Electrophysiol. 2013 Aug;24(8):875-81. doi: 10.1111/jce.12141. Epub 2013 Apr 11. PMID 23577826

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 44 patients were enrolled over 4 months; 6 patients withdrew: 4 patients had the device removed before study completion and 2 patients did not return for the required follow-up. The remaining 38 patients completed the study requirements and are reported in the final results.
Groups:
- CM and Reveal XT: This was the non-randomized phase of the study in the first six months of evaluation.
Period: 1 - 6 Months (Ron-randomized)
Arm/Group | Conventional Monitoring Strategy | Reveal XT | CM and Reveal XT
Started | 0 | 0 | 38
Completed | 0 | 0 | 38
Not Completed | 0 | 0 | 0
Period: 6 - 12 Months (Randomized)
Arm/Group | Conventional Monitoring Strategy | Reveal XT | CM and Reveal XT
Started | 18 | 20 | 0
Completed | 13 | 20 | 0
Not Completed | 5 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Monitoring Strategy | Reveal XT | Total
Number analyzed (Participants) | 18 | 20 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 11 | 22
  >=65 years | 7 | 9 | 16
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57 (12) | 61 (9) | 59.4 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 16 | 17 | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 18 | 20 | 0

OUTCOME MEASURES:

1. Primary Outcome: Arrhythmia Burden
Description: The primary outcome will be arrhythmia recurrences (atrial fibrillation and/or other atrial arrhythmias) after atrial fibrillation ablation over the initial 6 months and one year post-ablation as detected by the implantable loop recorder versus the conventional monitoring strategy. Months 1- 6 patients were being monitored by CM and ILR and in months 6 - 12 they were randomized to either ILR or CM.
Time Frame: 6 and 12 months
Population: Some participants withdrew before completing the full 1 year of required follow-up. In the first 6 months all 38 of the remaining patients arrhythmia recurrence was assessed using CM and Reveal XT. Participants were randomized in this phase to either CM or Reveal XT arms.
Measure: Count of Participants; unit: Participants
Groups:
- Reveal XT and Conventional Monitoring: This was the non-randomized phase of the study in the first six months of evaluation.
Arm/Group | Conventional Monitoring Strategy | Reveal XT | Reveal XT and Conventional Monitoring
Number analyzed (Participants) | 38 | 38 | 38
Participants
  First 6 months (non randomized) | 7 | 18 | 18
  6 -12 months (randomized): number analyzed (Participants) | 13 | 20 | 0
  6 -12 months (randomized) | 5 | 5 |

2. Secondary Outcome: Detection of Actionable Events Resulting in Change of Clinical Care
Description: Change of clinical care include initiation of previously discontinued and/or new anti-arrhythmic drugs, decision for repeat ablation, hospitalization for arrhythmias, discontinuation or reinitiation of atrio-ventricular nodal blocking agents, discontinuation or reinitiation af anticoagulation after ablation and/or decision to implant a pacemaker and/or defibrillator.
Time Frame: 12 months
Population: Participants were monitored for this end point regardless of the randomization strategy to ensure patient safety.
Measure: Count of Participants; unit: Participants
Groups:
- Reveal XT: Subjects will be monitored using the conventional monitoring strategy for the first 6 months post-ablation. During the next 6 months, subjects will be monitored using the data from the Reveal device, transmitted from home every 30 days.
  Reveal XT implantable loop recorder: All study participants will receive the Reveal XT implantable loop recorder immediately after completion of the ablation procedure.
  For details, please refer to the following citation of the published study: Kapa, et al, Journal of Cardiovascular Electrophysiology 2013; DOI:10.1111/JCE. 12141
Arm/Group | Conventional Monitoring Strategy | Reveal XT
Number analyzed (Participants) | 38 | 38
Participants | 0 | 5

ADVERSE EVENTS:
Arm/Group | Conventional Monitoring Strategy | Reveal XT
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/20
Other Adverse Events (participants affected / at risk) | 0/18 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No